CLINICAL TRIAL: NCT00415103
Title: AMENO-2: Fase IV Study, National, Multiple Centers, Competitive, Randomized, Double Blind, Controlled With Parallel Groups to Determinate the Security, Tolerability and Efficacy of Aprepitant Plus Palonosetron Versus Granisetron in the Prevention of Nausea and the Emesis Induced by Chemotherapy in Patients Treated With Haematopoietic Progenitors
Brief Title: AMENO-2: Aprepitant Plus Palonosetron Versus Granisetron in the Prevention of Nausea and the Emesis Induced by Chemotherapy in Patients Treated With Haematopoietic Progenitors
Acronym: AMENO-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Pethema, pethema
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-00055-18
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Leukemia; Lymphoma
Keywords: Emesis; Nausea; leukemia; lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Vomiting; Nausea | interventions — Aprepitant; Palonosetron; Granisetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Aprepitant: 125 mg oral day 1, follows by 80 mg oral every 24 hours in next days Palonosetrón: 0.25 mg iv every 48 horas starting day 1
  Interventions: Drug: Aprepitant; Drug: Palonosetron
- 2 (Active Comparator): Granisetrón : 3 mg iv day, all days the patient will be treated with chemotherapy, and Aprepitant placebo 125 mg oral, day 1, and 80 mg next days in chemotherapy treatment.
  Interventions: Drug: Granisetron

INTERVENTIONS:
Drug: Aprepitant — Aprepitant: 125 mg oral day 1, follows by 80 mg oral every 24 hours in next days
  Arms: 1
Drug: Palonosetron — Palonosetrón: 0.25 mg iv every 48 hours, starting day 1
  Arms: 1
Drug: Granisetron — Granisetrón : 3 mg iv day, all days the patient will be treated with chemotherapy, and Aprepitant placebo 125 mg oral, day 1, and 80 mg next days in chemotherapy treatment
  Arms: 2

SUMMARY:
The purpose of this trial is to determinate the security, tolerability and efficacy of aprepitant plus palonosetron versus granisetron in the prevention of nausea and emesis induced by chemotherapy in patients treated with haematopoietic progenitors transplant.

DETAILED DESCRIPTION:
Patients with haematopoietic cancer (as leukaemia and lymphomas) that are treated with high doses of intense chemotherapy for the haematopoietic progenitors transplant experiment intense nausea and emesis related to this chemotherapy treatment.

The introduction of regimens with antagonist of 5HT3 receptors (ondansetron, tropisetron, granisetron) seems to have reduced the magnitude of the problem in the first 24 hours after the beginning of the chemotherapy. However, in spite of the use of these drugs, it is very frequency to observe intense nausea and emesis induced by chemotherapy especially in the latest period (after 24 h).

MASCC guides establish that It is not possible to give firm recommendations in the prevention of the NVIQ for these patients. Currently, the treatment of this problem in patients that go through a total body irradiation is made with antagonist of 5HT3 receptors with or without Dexamethasone.

There is neither recommendation regarding the antiemetic prophylaxis in chemotherapy treatments with high emetogenic power of several days duration. However, there is controversy about the use of high doses of steroids to avoid the latest emesis in transplant patients ( because of the high doses of steroids, Its continuous use during several days in this clinical situation and because of the possible worsening of the immunodeficiency inherent to the oncohematology illness/the previous chemotherapy treatment received by the patient). In patients that go trough a haematopoietic progenitor's transplant, many teams prefer to avoid the use of steroids. Main clinical guides do not offer firm recommendations regarding antiemetic prophylaxis protocols in the TPH and antagonists of 5-HT3 receptors are commonly used in practice.

AMENO-1 study demonstrated that the incidence of NVIQ is high even with an anti-5HT3 daily prevention (experimenting vomits or requiring rescue treatment for 81% of the TPH receptors), this significantly ameliorated their quality of life.

Currently, there are new drugs with new action mechanisms and a probable synergy between them that increase control of the NVIQ out of the transplant field. For that reason we have designed a study with the purpose of evaluating whether these new drugs ameliorate the control that we currently have of NVIQ (which is far from optimal).

To avoid differences in terms of posology regimes, granisetron will be used as the common treatment with one daily dose of 3mg/day. The new experimental regime that we propose includes two newly commercialized drugs with complementary and different mechanisms of action that have demonstrated their efficacy and their security in the very emetogenic chemotherapy administrated only one day: aprepitant and palonosetron.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or up
* Will go through a Haematopoietic progenitors transplant (of mother cells from periphery blood or bone marrow with at least a 5 days long previous regime (with or without radiotherapy)
* women in fertile age must give negative in the pregnancy test in serum or in urine, sensible to 25 UI of β-hCG, in the visit before the study and accept to use a contraceptive double barrier method at least from the 14 previous days to the administration of the first dose of the study drug to the 14 following days after the last dose.
* Patient has a Karnofsky punctuation ≥60
* Patient has an life expectancy ≥1 month
* Patient is capable to read, understand and to complete the study questionnaires including the questions which require a visual analogy scale answer
* Patient understands the study procedure and agrees to participate in it, giving his written consent.
* Patient is going through one of these previous regimens:
* CBV (ciclofosfamide, BCNU and VP-16)
* BEAM (BCNU, VP-16, araC, melphalan)
* Regimens with BUCY (Busulfan x 4 days and ciclofosfamide with or without other agents)
* CYTBI (ciclofosfamide plus total body irradiation with/without others agents)

Exclusion Criteria:

* Patients that are in one of these situations if, according to investigator's opinion, it prevents their participation in the study.
* Mental disability or emotional or psychiatric significant disorder
* Patient consumes any kind of drug, included marijuana, or the investigator determines that he has excessive alcohol consumption.
* Patient has any kind of infection (e.g. pneumonia) or any other uncontrolled disease (e.g. digestive obstruction) different to the process that, in the investigator's opinion, could mix the study's results or put the patient at risk if the drug is administrated.
* Patient has history of hypersensitivity to granisetron, palonosetron or aprepitant.
* Patient has received any non proven drug (investigation) in the last 4 weeks.
* Patient has history or present history of cardiac conduction disorders specially QTC interval. Anti-arrhythmic use or electrolytic disorders capable of giving cardiac conduction disorders.
* Abnormal lab values
* AST >2.5 X superior limit of normality
* ALT >2.5 x superior limit of normality
* Bilirubin >1.5 x superior limit of normality
* Creatinine >1.5 x superior limit of normality
* Patients that in the 48 hours before day 1 of the study they have been treated with the following antiemetics:
* 5HT-3 antagonist (ondansetron, granisetron, dolasetron, or tropisetron)
* Fenotiacines
* Butyrophenones: (haloperidol or droperidol)
* Benzamides: metoclopramide or alizapride
* Domperidone
* Cannabinoids
* Patient who has started to receive treatment with benzodiazepines or with opioids in the first 48 hours before the day 1 of the study, except unique daily doses of triazolam, temazepam, lorazepam and midazolam. The continuation of the chronic treatment with benzodiazepins or with opioids is authorized as long as this treatment has been initiated at least 48 hours before day 1 of the study (considering that they can increase their levels.)
* Patient is taking or has taken in the 7 days before day 1 of the study the following substrates of the CYP3A4:
* Terfenadine
* Cisapride
* Astemizol
* Pimozide Or the following CYTP3A4 inhibitors
* clarithromycin : azithromycin, erythromicin aroxithromycin nd are allowed
* Ketoconazole or itraconazole (fluconazol is allowed)
* Patient is taking or has taken in the 30 days before day 1 of the study the following substrates of the CYP3A4:
* Barbiturics
* Rifampicin or rifabutin
* Carbamazepin or fenitoin. The administration of fenitoin as prophylaxis in regimens with busulfan of short duration is allowed in the following cases:

  * This is a common regimen of conditioning in the transplant:
  * The short time of treatment together -5 days maximum- and
  * With the recommendation to monitorize the levels of fenitoin (keeping in mind that the mutual interaction between aprepitant and fenitoin can decrease the level of both.)
* Patient is taking or has taken in the 7 days before day 1 of the study, steroids (They can be administrated as a rescue antiemetic if it is indicated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2006-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Determinate the security, tolerability and efficacy of aprepitant plus palonosetron versus granisetron in the prevention of nausea and emesis induced by chemotherapy in patients treated with haematopoietic progenitors transplant | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: López Javier, Dr, Study Chair — Hospital Universitario Ramon y Cajal
Locations (5):
- Spain (5):
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario la Princesa, Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander

REFERENCES:
- [Background] Bosi 1993; Agura 1995; Okamoto 1996
- [Background] MASCC Consensus Conference on Antihemetic Therapy, 2004)
- See also: Spanish association of Haematology — http://www.aehh.org